CLINICAL TRIAL: NCT03549195
Title: Novel Tumor Targeted Fluorescent Peptide TMTP1-ICG Mapping in Laparoscopic Sentinel Micro-metastasis Lymph Node Detection in Cervical Cancer Patients
Brief Title: TMTP1 Targeting Micro-metastasis LN in Laparoscopic SLN Detection in Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ding Ma, Director, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMTP1-ICG-03
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Cervical Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ICG (Active Comparator)
  Interventions: Procedure: ICG
- ICG-CP (Active Comparator): CP, control peptide
  Interventions: Procedure: ICG-CP
- ICG-TMTP1 (Experimental): also named as TMTP1-ICG
  Interventions: Procedure: ICG-TMTP1

INTERVENTIONS:
Procedure: ICG — The ICG powder was diluted and injected into the cervix, divided into 3 and 9 o'clock position, 4 hours before surgery.
  Arms: ICG
Procedure: ICG-CP — The ICG-CP powder was diluted and injected into the cervix, divided into 3 and 9 o'clock position, 4 hours before surgery.
  Arms: ICG-CP
Procedure: ICG-TMTP1 — The ICG-TMTP1 powder was diluted and injected into the cervix, divided into 3 and 9 o'clock position, 4 hours before surgery.
  Arms: ICG-TMTP1

SUMMARY:
Investigators aimed to determine the validity of the investigator's novel tumor targeted fluorescent peptide TMTP1-ICG to increased accuracy of laparoscopic SLN mapping

ELIGIBILITY:
Inclusion Criteria:

* Without childbearing requirements at the time of consent.
* FIGO stage IB1, IIA1 cervical cancer and is a candidate for laparoscopy intervention, with lymph node dissection being a part of the surgical plan.
* Subject has provided written informed consent.

Exclusion Criteria:

* Breast-feeding or pregnant.
* Ongoing participation in another clinical trial with an investigational drug with 3 months
* Own allergy towards ICG and/or alcohol
* Diagnosis of bacterial vaginosis, fungal vaginitis, sexually transmitted diseases
* Patients with cardiac dysfunction or hepatic insufficiency or renal insufficiency

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection rate of micro-metastasis sentinel lymph node | 7 days
  Detection of micro-metastasis sentinel lymph node per patient

SECONDARY OUTCOMES:
Sensitivity | 7 days
  Sensitivity of SLN mapping of TMTP1-ICG compared to the sensitivity of SLN mapping of ICG or ICG-CP
Specificity | 7 days
  Specificity of SLN mapping of TMTP1-ICG compared to the sensitivity of SLN mapping of ICG or ICG-CP
Incidence of adverse events | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, HUST, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No